CLINICAL TRIAL: NCT07115706
Title: A Multi-center Prospective Observational Study to Evaluate the Effectiveness and Safety of JAQBO® Tab. 20 mg(Zastaprazan Citrate) in Erosive Gastroesophageal Reflux Disease
Brief Title: JAQBO® Tab. 20 mg(Zastaprazan Citrate) in Erosive GERD
Status: Not yet recruiting | Type: Observational
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JL-JAQ-403
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Erosive Gastroesophageal Reflux Disease
Keywords: Erosive Gastroesophageal Reflux Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group1: those with a condition

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of JAQBO® Tab. 20 mg(Zastaprazan citrate) patients who have been prescribed the investigational drug.

DETAILED DESCRIPTION:
Multi-center prospective observational study

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 19 years or older who have been diagnosed with erosive reflux disease (ERD)
* subjects who have voluntarily decided to participate in this observational study and have provided written informed consent after receiving the study information and consent form

Exclusion Criteria:

* Subjects who fall under the contraindications listed in the precautions for use section of the approved labeling for Fexuclu tablets:

  1. Subjects with hypersensitivity or a history of hypersensitivity to the investigational drug or any of its components
  2. Subjects currently taking medications containing atazanavir, nelfinavir, or rilpivirine
  3. Pregnant women, women who may be pregnant, or breastfeeding women
  4. Subjects with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Subjects deemed inappropriate for participation in the study at the investigator's discretion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital
Sampling Method: Probability Sample
Enrollment: 7150 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Reflux Disease Questionnaire (RDQ) at Week 8 | Week 8
  This questionnaire is a self-reported instrument designed to assess the main symptoms of gastroesophageal reflux disease (GERD), including heartburn, acid regurgitation, and dyspepsia. It consists of a total of 12 items, each evaluating the frequency and severity of symptoms using a 6-point scale (0 to 5). In this observational study, only heartburn and acid regurgitation symptoms are assessed. The questionnaire is completed by the study participants themselves, and higher total scores indicate more severe symptoms.

IPD SHARING:
Plan to Share IPD: Undecided